CLINICAL TRIAL: NCT05947994
Title: Elucidate Outcomes of Elective High-grade/Total Occlusion Intracranial Arteries Using Low-profile Self-expanding Stent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Can Tho Stroke International Services Hospital (Other)
Collaborators: Acandis GmbH (Industry)
Responsible Party: Principal Investigator, Dr. Cuong Tran Chi, Director - Doctor, Can Tho Stroke International Services Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CRESIS
Record Dates: First submitted 2023-07-09; First posted 2023-07-17 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Intracranial Atherosclerosis; Stent Stenosis; Ischemic Stroke
Keywords: Ischemic stroke; Intracranial Atherosclerosis; Intracranial stenting
MeSH Terms: conditions — Intracranial Arteriosclerosis; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Optimal medical therapy failure (Experimental): Symptomatic ischemic stroke patients were treated with Credo® Stent
  Interventions: Procedure: Intracranial stenting with Credo® stent

INTERVENTIONS:
Procedure: Intracranial stenting with Credo® stent — Symptomatic ischemic stroke patients were treated with Credo® Stent

SUMMARY:
Intracranial atherosclerotic disease (ICAD) is a high prevalent cause of stroke, especially in Asian population and can be categorized as either symptomatic (resulting in acute ischemic stroke) or asymptomatic. Treatment for patients who failed with optimal medical therapy (OMT) is still elucidating.

DETAILED DESCRIPTION:
In symptomatic ischemic stroke due to intracranial large severe stenosis or occlusive artery, the choice for treatment has remained controversial after results of the Stenting versus Aggressive Medical Therapy for Intracranial Arterial Stenosis (SAMMPRIS) trial because it demonstrated that the efficacy of medical treatment was superior to intracranial stenting (IS) in the low risk of periprocedural stroke or death. However, this conclusion has influenced the role of IS in the secondary prevention of ischemic stroke and recovery time for a long time because of the improper patient selection of this trial such as no evidence of medical failure, IS in case of moderate intracranial stenosis and IS in patients with transient ischemic attacks only. Recently, the Food and Drug Administration (FDA) mandated study about IS, the Wingspan Stent System Post Market Surveillance (WEAVE) trial, reported not only 97.4% patients with no complication at 72 hours, but also a relatively low 8.5% recurrent stroke and death rate during 1 year in the Wingspan One Year Vascular Imaging Events and Neurologic Outcomes (WOVEN) study about Wingspan stent (Stryker, Kalamazoo, MI). In case of the symptomatic stenosis greater than 70%, the probability of recurrent stroke and transient ischemic attack in the territory of the symptomatic stenotic artery in 1 year was 23% and 14%, respectively, despite treatment with antithrombotic therapy and standard management of vascular risk. Given a lot of patients with symptomatic ischemic stroke who have some adjustable indications for intracranial stenting deployment with Wingspan stent in the world and a paucity of evidence from the comprehensive stroke centers about other self-expanding stents, Credo stent (Acandis GmbH, Pforzheim, Germany), our purpose was to compare the periprocedural complication and rate of 1-year recurrent ischemic stroke associating to the IS between beyond 7 days from acute stage and the progressive ischemic stroke time.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of severe intracranial stenosis
* Target intracranial artery ≥ 2 mm
* Absence of intracranial hemorrhage
* Procedure treated with the Credo stent (Acandis, Pforzheim, Germany)

Exclusion Criteria:

* Premorbid modified Rankin Scale (mRS) score ≥ 2
* Intracranial rescue stenting for acute ischemic stroke within 24 hours
* Loss to follow-up after discharge
* Systemic lupus erythematosus
* More procedures at the same time

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-04-20 (Actual)

PRIMARY OUTCOMES:
Rate of the critical adverse events | After procedure within 24 hours
  The critical adverse events: intracranial hemorrhage, new infarct
Rate of 1-year recurrent ischemic stroke | During 1 year after procedure
  Rate of 1-year recurrent ischemic stroke in the territory of the symptomatic intracranial artery

CONTACTS AND LOCATIONS:
Overall Officials: Cuong C Tran, PhD, Principal Investigator — Can Tho Stroke International Services General Hospital
Locations (1):
- Can Tho Stroke International Service General Hospital, Can Tho, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alexander MJ, Zauner A, Gupta R, Alshekhlee A, Fraser JF, Toth G, Given C, Mackenzie L, Kott B, Hassan AE, Shownkeen H, Baxter BW, Callison RC, Yu W. The WOVEN trial: Wingspan One-year Vascular Events and Neurologic Outcomes. J Neurointerv Surg. 2021 Apr;13(4):307-310. doi: 10.1136/neurintsurg-2020-016208. Epub 2020 Jun 19. PMID 32561658
- [Background] Alexander MJ, Zauner A, Chaloupka JC, Baxter B, Callison RC, Gupta R, Song SS, Yu W; WEAVE Trial Sites and Interventionalists. WEAVE Trial: Final Results in 152 On-Label Patients. Stroke. 2019 Apr;50(4):889-894. doi: 10.1161/STROKEAHA.118.023996. PMID 31125298
- [Background] Tran CC, Le MT, Baxter BW, Nguyen-Luu G, Ngo MT, Nguyen-Dao NH, Duong-Hoang L, Mai-Van M, Nguyen MD. Rescue intracranial stenting in acute ischemic stroke: a preliminary Vietnamese study. Eur Rev Med Pharmacol Sci. 2022 Oct;26(19):6944-6952. doi: 10.26355/eurrev_202210_29875. PMID 36263574
- [Background] Le MT, Tran CC, Nguyen-Luu G, Ngo MT, Nguyen-Dao NH, Duong-Hoang L, Mai-Van M, Nguyen MD. Rescue stenting after the failure of intravenous thrombolysis and bridging thrombolysis: an initial Vietnamese report. Eur Rev Med Pharmacol Sci. 2022 Dec;26(24):9162-9169. doi: 10.26355/eurrev_202212_30667. PMID 36591828